CLINICAL TRIAL: NCT06625437
Title: Evaluation of the Effectiveness of Acceptance and Commitment Therapy for General Mental Health Concerns in HIV-Positive Men
Brief Title: ACT for HIV-Positive Men
Acronym: ACT for HIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nicholas C. Borgogna, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300013506; Start-up (Other: UAB)
Record Dates: First submitted 2024-09-26; First posted 2024-10-03 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Stress; Anxiety; Mental Disorder; Distress-based Psychopathology
MeSH Terms: conditions — Anxiety Disorders; Mental Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Pre-post design with single group of participants who will each receive the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acceptance and commitment therapy (Experimental): Trial of acceptance and commitment therapy for hiv-positive men.
  Interventions: Behavioral: Acceptance and commitment therapy

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy — Acceptance and commitment therapy is a psychotherapy focused at increasing psychological flexibility and an individual's engagement in valued activities rather than focusing solely or primarily on reducing psychiatric symptoms

SUMMARY:
The purpose of the current study is to examine the feasibility and effectiveness of acceptance and commitment therapy, a specific form of cognitive-behavioral therapy, for treating general mental health concerns among HIV-positive men.

DETAILED DESCRIPTION:
The purpose of the current study is to examine the feasibility and effectiveness of acceptance and commitment therapy, a specific form of cognitive-behavioral therapy, for treating general mental health concerns among HIV-positive men.

ELIGIBILITY:
Inclusion Criteria:

* identify as a man
* be at least 18 years old
* has been diagnosed with HIV by a healthcare professional

Exclusion Criteria:

* has engaged in self-harm within the last three months
* has attempted suicide within the last year
* has had an active plan to attempt suicide within the last 30 days
* is currently diagnosed with any eating disorder
* has experienced hallucinations or delusions within the last 30 days
* has used narcotics within the last 7 days (heroin, meth, crack cocaine, opioids)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 24 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 Screener | Administered at baseline and immediately after final intervention session (8th/final session; each session is 1 hour)
  Measure of depressive symptoms
PTSD Checklist-5 | Administered at baseline and immediately after final intervention session (8th/final session; each session is 1 hour)
  Measure of post-traumatic stress symptoms
Yale-Brown Obsessive Compulsive Scale | Administered at baseline and immediately after final intervention session (8th/final session; each session is 1 hour)
  Measure of obsessive-compulsive disorder symptoms
Alcohol Use Disorders Identification Test | Administered at baseline and immediately after final intervention session (8th/final session; each session is 1 hour)
  Measure of alcohol use
HIV stigma scale | Administered at baseline and immediately after final intervention session (8th/final session; each session is 1 hour)
  Measure of facets of stigma experienced by individuals with HIV
Internalized homophobia scale | Administered at baseline and immediately after final intervention session (8th/final session; each session is 1 hour)
  Measure of internalized homophobia
Brief pornography screen | Administered at baseline and immediately after final intervention session (8th/final session; each session is 1 hour)
  Measure of concerning pornography use
Life Quality Scale | Administered at baseline and immediately after final intervention session (8th/final session; each session is 1 hour)
  Measure of life quality
Experiential Avoidance Rating Scale | Administered at baseline, every two weeks (every second therapy session) during intervention, and immediately after final intervention session (8th/final session; each session is 1 hour)
  Measure of experiential avoidance
National Institute of Drug Abuse Modified Alcohol, Smoking, and Substance Involvement Screening Test | Administered at baseline and immediately after final intervention session (8th/final session; each session is 1 hour)
  Measure of drug use
High risk sexual behaviors | Administered at baseline and immediately after final intervention session (8th/final session; each session is 1 hour)
  * Frequency of sex with penetration
  * Frequency of condom use
  * Frequency of oral sex
  * Frequency of sexual partners
Generalized Anxiety Disorder-7 Screener | Administered at baseline and immediately after final intervention session (8th/final session; each session is 1 hour)
  Measure of anxiety symptoms
PSYFLEX | Administered at baseline, every two weeks (every second therapy session) during intervention, and immediately after final intervention session (8th/final session; each session is 1 hour)
  Measure of psychological flexibility

SECONDARY OUTCOMES:
Therapeutic Alliance Scale | Administered immediately after final intervention session (8th/final session; each session is 1 hour)
  Measure of patient and therapist alliance

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Borgogna, PhD, Principal Investigator — University of Alabama at Birmingham; Drew Whittington, MS, MA, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Dataset will be shared with requesting researchers
Time Frame: When results are published
Access Criteria: Requesting researchers